CLINICAL TRIAL: NCT01368562
Title: A Compassionate Use Study of Methylnaltrexone in Patients With Opioid-Induced Side Effects
Brief Title: Compassionate Use Study of Methylnaltrexone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 901
Expanded Access: Available
Record Dates: First submitted 2011-05-27; First posted 2011-06-08 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Opioid-induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylnaltrexone (Experimental): Participants will receive single dose of MNTX 0.15 milligrams per kilogram (mg/kg) subcutaneously (SC). Subsequent dosing could be adjusted upward (to a maximum of 0.3 mg/kg) to achieve a desired clinical response or decreased to improve tolerability.
  Interventions: Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Methylnaltrexone — Methylnaltrexone will be administered as per the dose and schedule specified in the arm.

SUMMARY:
This is an open label compassionate use study of subcutaneously administered methylnaltrexone (MNTX) in participants with advance medical illness and opioid-induced constipation.

ELIGIBILITY:
Inclusion Criteria:

* Advanced medical illness (that is; terminal illness, such as incurable cancer or end stage aqcuired immunodeficiency syndrome [AIDS]) with a life expectancy of one to six months.
* On an opioid regimen for the control of pain/discomfort for at least seven days.
* Has opioid-induced constipation.
* Stable vital signs and systolic blood pressure greater than or equal to (>=) 85 millimeters of mercury (mmHg), and diastolic blood pressure >=45 mmHg (Supine or sitting).
* Females of childbearing potential must have a negative pregnancy test (serum or urine).
* On a laxative regimen (for example, stool softener and SENNA or equivalent) for at least 3 days prior to treatment. Participants who have discontinued laxatives due to intolerability or lack of efficacy are also eligible.

Exclusion Criteria:

* Participants with known hypersensitivity to methylnaltrexone, naltrexone or naloxone.
* Participants who received any investigational new drug (experimental) except for methylnaltrexone in the previous 30 days.
* Participants who are constipated with a disease process suggestive of gastrointestinal obstruction, impaction or diagnosed with a current abdominal pathologic process which may represent a non-opioid cause of bowel dysfunction.
* Participants who are constipated and have active, clinically significant diverticulitis.
* Participants with a surgically acute abdomen.
* Participants being treated with opioids for diarrhea, dyspnea, cough, pulmonary edema, or congestive heart failure.
* Individuals with a known drug addiction.
* Females who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-01-24 (Actual); Primary Completion 2008-06-02 (Actual); Study Completion 2008-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Companies
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylnaltrexone: Participants received single dose of methylnaltrexone (MNTX) 0.15 milligrams per kilogram (mg/kg) subcutaneously (SC) initially. Subsequent dosing was adjusted upward (to a maximum of 0.3 mg/kg) to achieve a desired clinical response or decreased to improve tolerability. Median treatment duration was 25 days.
Period: Overall Study
Arm/Group | Methylnaltrexone
Started | 26
Received at Least 1 Dose of Study Drug | 25
Completed | 7
Not Completed | 19
Not completed — Adverse Event | 1
Not completed — Disease progression | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 6
Not completed — Unresponsive to treatment | 5
Not completed — Other | 3
Not completed — Other than specified | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who provided a signed and dated written informed consent form (ICF).
Groups:
- Methylnaltrexone: Participants received single dose of MNTX 0.15 mg/kg SC initially. Subsequent dosing was adjusted upward (to a maximum of 0.3 mg/kg) to achieve a desired clinical response or decreased to improve tolerability. Median treatment duration was 25 days.
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Mean age data of safety evaluable participants (all enrolled participants who received at least one dose of study drug) was calculated and reported.
  years
    number analyzed (Participants) | 25
    (all) | 59.4 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 24
  Hispanic | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Opioid Induced Side Effects
Description: Opioid induced side effects included nausea, myoclonus, mental clouding (confusional state), vomiting, sedation, pruritus, sweating (hyperhidrosis), constipation, and urinary retention. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From start of treatment until end of study (up to maximum 3.4 years)
Population: All enrolled participants who provided a signed and dated written ICF.
Measure: Count of Participants; unit: Participants
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 26
Participants
  Nausea | 3
  Myoclonus | 1
  Vomiting | 3
  Sedation | 1
  Constipation | 1
  Urinary retention | 3
  Mental clouding | 4
  Sweating | 2
  Pruritus | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until end of study (up to maximum 3.4 years)
Description: Safety evaluable participants included all enrolled participants who received at least one dose of study drug.
Arm/Group | Methylnaltrexone
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone (N=25)
Small intestinal obstruction (Gastrointestinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Asthenia (General disorders) | 1
Pain (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Convulsion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone (N=25)
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dizziness (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Bronchitis bacterial (Infections and infestations) | 1
Abdominal distension (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Oedema peripheral (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Faecaloma (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Urinary tract infection (Infections and infestations) | 2
Sedation (Infections and infestations) | 1
Haematuria (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Yawning (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Lacrimation increased (Eye disorders) | 1
Catheter related complication (General disorders) | 1
Chest discomfort (General disorders) | 1
Secretion discharge (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Feeling abnormal (General disorders) | 1
Fatigue (General disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Oral intake reduced (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 2
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Creatinine renal clearance decreased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Cyanosis (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Pallor (Vascular disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Asthenia (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.